CLINICAL TRIAL: NCT03039244
Title: Evaluation of Antimicrobial Photodynamic Therapy in Multiples Episodes as an Adjunct to Non-surgical Periodontal Treatment in Smokers
Brief Title: Evaluation of Antimicrobial Photodynamic Therapy as an Adjunct to Periodontal Treatment in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Vice-Director of School of Dentistry of Ribeirão Preto, University of São Paulo, Brazil, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36933014.4.0000.5419
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Chronic Periodontitis
Keywords: Photochemotherapy; Photosensitizing agents; Smokers
MeSH Terms: conditions — Chronic Periodontitis | interventions — Photochemotherapy; Laser Therapy; Control Groups; Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: The study type will be split mouth with two pairs of contralateral uni-root teeth with proximal periodontal sites presenting probing depth ≥ 5 mm for the clinical, microbiological and immunological assessment. A random number table will be generated by a computer program, each of the selected pairs dental receive the following treatments: SRP or SRP + several aPDT episodes
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A random number table will be generated by a computer program, each of the selected pairs dental receive the following treatments: SRP or SRP + several aPDT episodes. The clinical, immunological and microbiological parameters will be evaluated at baseline (pre-intervention) and after the completion of non-surgical periodontal therapy. The periodontal clinical examinations (pre and post-intervention) will be performed by a single trained and calibrated examiner, who unknown the experimental groups of this study. Examiners are also blind to study the immunological and microbiological analyzes. SRP procedures and use of the aPDT protocol should be performed by other trained operator for these purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): After Scaling and root planing, periodontal pockets will receive the antimicrobial (aPDT) photodynamic therapy. Shortly phenothiazine hydrochloride photosensitizing is applied at a concentration of 10mg/mL from the pocket bottom to the gingival margin. After 1 minute, irrigation is performed from periodontal pockets with distilled water to remove excess dye. The stained area is then irradiated with a diode laser with 660 nm of wavelength and maximum power of 60 mW/cm², through a fiber-optic probe of 0.6 mm diameter. Exposure to radiation will occur at six sites per tooth under treatment, making the total time of 1 minute per element, or the equivalent of 10 seconds per site. The aPDT applications will be repeated in the same way until the second week in the days 2, 7 and 14.
  Interventions: Other: Photodynamic therapy; Device: Diode Laser
- Control Group (Sham Comparator): A sham procedure will be held simultaneously in pairs of contralateral teeth selected that will not receive the aPDT (control group).
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Photodynamic therapy — After Scaling and root planing, periodontal pockets will receive the antimicrobial (aPDT) photodynamic therapy. Shortly phenothiazine hydrochloride photosensitizing is applied at a concentration of 10mg/mL from the pocket bottom to the gingival margin. After 1 minute, irrigation is performed from periodontal pockets with distilled water to remove excess dye. The stained area is then irradiated with a diode laser with 660 nm of wavelength and maximum power of 60 mW/cm², through a fiber-optic probe of 0.6 mm diameter. Exposure to radiation will occur at six sites per tooth under treatment, making the total time of 1 minute per element, or the equivalent of 10 seconds per site. The aPDT applications will be repeated in the same way until the second week in the days 2, 7 and 14.
  Other Names: Laser therapy
  Arms: Test Group
Other: Control Group — A sham procedure will be held simultaneously in pairs of contralateral teeth selected that will not receive the aPDT (control group).
  Other Names: Sham procedure
  Arms: Control Group
Device: Diode Laser
  Arms: Test Group

SUMMARY:
The study proposes to assess the effect of multiple applications of antimicrobial Photodynamic Therapy (aPDT) as an adjunct to non-surgical periodontal treatment (nsPT) in smokers without use of antibiotics. Twenty smokers with a clinical diagnosis of chronic periodontitis will be treated in a split-mouth design study to either aPDT associated with scaling and root planing (SRP) or SRP only. aPDT will be performed by using a laser light source with 690 nm wavelength associated with a phenothiazine photosensitizer. The applications will occur in four episodes (at days 0, 2, 7 and 14). All patients will be monitored for 90 days. Plaque index, probing depth, clinical attachment level and bleeding on probing will be performed at baseline (pre-intervention period) and 30 and 90 days after the (nsPT). Subgingival plaque samples will be collected (at baseline and 30 and 90 days after the nsPT) and the counts of 40 subgingival species will be determined using DNA-DNA checkerboard hybridization. Gingival crevicular fluid samples will be collected (at Day 0, 14, 30 and 90 after the nsPT) and the levels of Interleukin 1 beta, Interleukin 10 and Tumor Necrosis Factor alpha (Luminex) will be evaluated. Salivary cotinine levels will also be evaluated at baseline. Data obtained will be statistically analyzed.

DETAILED DESCRIPTION:
MATERIALS AND METHODS

Consent to search - All patients will receive detailed information about experiment (goals, benefits, risks and discomforts) in accordance with a consent form in this research. All procedures will be subject to approval of the Ethics Committee (CEP) of Ribeirão Preto Dental School (FORP), University of São Paulo (USP).

Sample Size Calculation - The sample size was determined to provide 80% power to recognize a significant difference of 1 mm (d) between groups with a 95% confidence interval (a = 0.05) and standard deviation (s) of 1.0 mm. Considering the changes in mean clinical attachment level (CAL) as the primary outcome variable and [Za (1.96) + Zb (0.84)]2 = 7.84. Size calculation was based on the following formula: n = {2[(s)2/(d)2]} · (Za + Zb)2. Therefore, a total of 16 patients were required. However, the number of patients enrolled in this study was 20, considering that some patients could be lost during follow-up.

Experimental Design -The selected subjects will receive specific oral hygiene instruction and supragingival scaling in all teeth, seven days before the start of interventions. The study type will be split mouth with two pairs of contralateral uni-root teeth with proximal periodontal sites presenting probing depth ≥ 5 mm for the clinical, microbiological and immunological assessment. A random number table will be generated by a computer program, each of the selected pairs dental receive the following treatments: SRP or SRP + several aPDT episodes. The clinical, immunological and microbiological parameters will be evaluated at baseline (pre-intervention) and after the completion of non-surgical periodontal therapy. The periodontal clinical examinations (pre and post-intervention) will be performed by a single trained and calibrated examiner, who unknown the experimental groups of this study. Examiners are also blind to study the immunological and microbiological analyzes. SRP procedures and use of the aPDT protocol should be performed by other trained operator for these purposes.

An impression with alginate will be performed in each patient to obtain the models of the dental arches and development of a guide plate on acetate with reference grooves to standardize the insertion and inclination of computerized periodontal probe (Florida Probe System, Florida Probe Corporation , Gainesville, FL, USA). The visible plaque index of each patient, will be assessed dichotomously (O'Leary et al., 1972) and determined by the percentage of tooth surfaces with plaque. In 6 sites of each tooth (mesio-buccal, buccal, distobuccal, mesio- lingual, lingual and disto-lingual) will be assessed clinical periodontal parameters: Probing Depth (mm) that will be measured from the gingival margin to the pocket bottom; relative Clinical Attachment Level (mm) that will be measured from the occlusal plate guide to the pocket bottom; Bleeding on probing, rated dichotomously (Ainamo, Bay, 1976), the presence of bleeding is considered positive when presented within 20s after the probe insertion for measuring probing depth. These clinical parameters and each patient's plaque index will be recorded at baseline (pre-intervention period) as well as +30 and +90 days after the non-surgical periodontal therapy.

Examiner Calibration - The Kappa index will be used to evaluate the examiner calibration for collection of clinical periodontal parameters in order to measure the intra-examiner agreement. According to the World Health Organization (WHO) for diagnostic criteria, acceptable index Kappa agreement must be greater or equal to 0.85 (WHO, 1997). This agreement level will be used for calibration of the examiner in this project. Ten patients will be selected, at least two pairs of contralateral teeth uni-roots with probe depth ≥5 mm in the proximal sites. Each patient is scanned twice using computerized periodontal probe (Probe Corporation Florida, Gainesville, FL, USA) with a 48-hour interval between the first and second examination in order to obtain the intra-examiner reliability, which will be measured by determining the Kappa index.

Immunologic Analysis - At baseline and on days +14, +30 and +90, after non-surgical periodontal therapy will be collected GCF samples from selected teeth. The supragingival plaque these elements will be removed and the sites will be gently dried with air jets and subsequently isolated using sterile cotton rolls. The GCF samples are obtained from the mesial and distal sites to the use of Periopaper strips (Oralflow Inc., Amityville, NY, USA). The strips will be carefully placed on the margin of the gingival sulcus for 30 seconds. The amount of absorbed gingival fluid will be determined by an electronic meter of wet mass Periotron (Oralflow Inc., Amityville, NY). The strips are placed in sterile eppendorf vials of the type which will be stored at a temperature of 80C for later quantification of cytokines (pg/ml) TNF-α, IL-1β and IL-10. Cytokine levels are determined using a 3-plex kit Millipore (Millipore Corporation, Billerica, MA, USA) 100TM and the Luminex system (Luminex, MiraiBio, Alameda, CA, USA).

Salivary Cotinine analysis - Cotinine is a metabolite of nicotine which allows monitoring patient exposure to nicotine (McGuire et al., 1989). Cotinine levels will be identified at baseline by immunoenzymatic analysis (ELISA) (Salimetrics Inc., State College, PA, USA) using a kit for the quantitative analysis of cotinine in saliva according to the manufacturer's instructions.

Microbiological Analysis - At baseline and on days +30 and +90, after performing non-surgical periodontal therapy, subgingival plaque samples of the selected teeth will be collected at the proximal periodontal pockets (mesial and distal). Counts of 40 subgingival species will be determined in each sample using the method checkerboard DNA-DNA hybridization (Birth et al., 2008). For the collection of subgingival plaque, the sites will be isolated with sterile cotton rollers and dry with air jets. The supragingival plaque will be removed carefully using a sterile curette. Subsequently, another sterile curette is used to collect subgingival plaque, starting from the deepest portion of the pocket to the coronal region. The samples will be transported in sterile Eppendorf vials and processing in Dental Molecular Diagnostics Laboratory of the School of Dentistry of Ribeirão Preto-USP

Non-surgical Periodontal Therapy - At 7 day prior to the non-surgical periodontal therapy all patients will pefrom a complete periapical radiographic examination of the entire mouth. They will be grouped into an oral hygiene program (OHP) according to the specific needs. In this program patients will receive instructions for effective self-plaque, including information about Bass technique (Bass, 1954) and interproximal cleaning with dental floss and interdental brushes. They will also be encouraged to brush the tongue once a day and receive a single dentifrice to be used during the whole experimental period (Colgate Total, Anakol Ind. Com. Ltda - Kolynos do Brasil - Colgate Palmolive Co., São Bernardo do Campo, SP, Brasil). After the completion of this oral hygiene program, patients will be submitted to evaluation of clinical periodontal parameters previously described, and also will be collected subgingival plaque and GCF samples on selected sites (baseline - pre-intervention period). Soon after, will receiving supragingival scaling and polishing with a coronary rubber cups in all teeth in the oral cavity.

Non-surgical periodontal therapy is initiated 7 days after the execution of the OHP and initial supragingival scaling. The treatment will be made by one skilled in Periodontology, at an interval of 24 hours by scaling (supragingival and subgingival) and root planing of all teeth with periodontal disease, using hand (Curetas Gracey, Hu-Friedy, Chicago, IL, EUA) and ultrasonic tools. The instrumentation will be held quadrant by quadrant, until adequate cleaning of the area and root planing, which will be checked with the help of an explorer. Individuals will receive professional cleaning biweekly up to three months after the end of nonsurgical periodontal therapy. In Fortnightly control and evaluation, patient cooperation towards the study will be monitored, verifying the state of oral hygiene.

Statistical Analysis - Normality and homoscedasticity of the data will be checked. The inter- and intra-group comparisons in different time intervals will be achieved through adequate parametric or non-parametric tests. For all statistical analysis will use a 5% significance level. All calculations are performed using SPSS software (SPSS, Chicago IL, EUA).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic periodontitis according to the international classification of periodontal diseases adopted by the American Academy of Periodontology (Armitage, 1999)
* periodontal pockets ≥ 5 mm
* smoking ≥ 20 cigarettes per day

Exclusion Criteria:

* Positive history of antibiotic therapy in the last six months
* Positive history of basic periodontal treatment in the last six months
* Involvement systemic that might interfere in disease progression or treatment response (eg .: diabetes, immune disorders)
* Pregnant
* Patients with extensive prosthetic wrap
* Patients with the need for antibiotic prophylaxis for performing routine dental procedures

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical Parameter | 2 years
  clinical attachment level of the selected periodontal sites

SECONDARY OUTCOMES:
Immunologic Analysis of the selected periodontal sites | 3 years
  Cytokine levels
Microbiological Analysis of the selected periodontal sites | 3 years
  periodontal pathogens counts
Salivary Cotinine analysis | 3 years
  cotinine levels
Clinical Parameter 2 | 2 years
  probing depth

CONTACTS AND LOCATIONS:
Locations (1):
- Mariana Sales, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Melo Soares MS, D'Almeida Borges C, de Mendonca Invernici M, Frantz FG, de Figueiredo LC, de Souza SLS, Taba M Jr, Messora MR, Novaes AB Jr. Antimicrobial photodynamic therapy as adjunct to non-surgical periodontal treatment in smokers: a randomized clinical trial. Clin Oral Investig. 2019 Aug;23(8):3173-3182. doi: 10.1007/s00784-018-2740-3. Epub 2018 Nov 3. PMID 30392080